CLINICAL TRIAL: NCT02087891
Title: Stress Free Now in a Corporate Call Center
Acronym: SFN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 11-254
Record Dates: First submitted 2014-02-26; First posted 2014-03-14 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CTL (No Intervention): Wait-list control, no intervention. Intervention offered after week 16 and outcomes are collected.
- Web-based stress management (WSM) (Experimental): Subjects randomized to this group will receive access to the WSM program to complete on their own time.
  Interventions: Behavioral: Web-based Stress Management Program (WSM)
- WSMg1 (Experimental): Subjects randomized to this group will receive access to WSM with group support. They will meet once per week for 1 hour. Meeting will be led by one of their peers who is a non-expert facilitator.
  Interventions: Behavioral: Web-based Stress Management Program (WSM); Behavioral: Group Support (WSMg1)
- WSMg2 (Experimental): Subjects randomized to this group will receive access to WSM and group support and clinical expert support. They will attend 4 weekly support groups led by a peer non-expert facilitator and 4 weekly support groups led by a clinical psychologist.
  Interventions: Behavioral: Web-based Stress Management Program (WSM); Behavioral: Group Support (WSMg1); Behavioral: Clinical Expert Support (WSMg2)

INTERVENTIONS:
Behavioral: Web-based Stress Management Program (WSM) — The intervention, developed by the Cleveland Clinic, is an 8-week online, interactive, educational program based on mindfulness meditation. Briefly, each week subjects are introduced to the (1) weekly audio introduction to the mindfulness theme or particular meditation technique of the week, (2) weekly audio meditation techniques for relaxation, (3) daily articles providing scientific evidence and merits of meditation, and (4) bi-weekly email reminders. The introductory talks and meditation exercises were also provided on compact discs (CD) in mp3 format.
  Other Names: Stress Free Now
  Arms: WSMg1; WSMg2; Web-based stress management (WSM)
Behavioral: Group Support (WSMg1) — Subjects will meet once per week for 1 hour during the 8-week duration and practice 2-minutes of deep breathing exercises, listen to 10-minutes audio recording of the weekly lesson and practice 20-30 minutes guided meditation exercise. The remainder of the time will be used to foster sharing experiences and answering specific questions related to the weekly lesson.
  Arms: WSMg1; WSMg2
Behavioral: Clinical Expert Support (WSMg2) — A clinical psychologist will replace the non-expert facilitator during 4 group support sessions.
  Arms: WSMg2

SUMMARY:
Psychosocial stress increases the risk for a multitude of diseases, including obesity, hypertension, and cardiovascular disease. Stress may also result in increased utilization of health care services. In the workplace, stress leads to emotional exhaustion, job dissatisfaction, lower productivity and impaired performance. Stress management programs and those based on mindfulness meditation have gained popularity in recent years. The purpose of this study is to evaluate the feasibility of an 8-week web-based mindfulness stress reduction program and its effectiveness in reducing work related stress and improving well-being in a large corporate call center.

ELIGIBILITY:
Inclusion Criteria:

* Frontline employee of large corporate call center
* Internet access

Exclusion Criteria:

* Manager or supervisor of large corporate call center

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Assess whether an 8-week mindfulness stress reduction online program is effective in improving mindfulness. | 8 weeks
  Outcome measured using Mindful Attention Awareness Scale (MAAS) questionnaire.
Assess whether an 8-week mindfulness stress reduction online program is effective in reducing stress mindfulness. | 8 weeks
  Outcome measured using the Perceived Stress Scale (PSS10) questionnaire.
Assess whether an 8-week mindfulness stress reduction online program is effective in decreasing burnout mindfulness. | 8 weeks
  Outcome measured using the Maslach Burnout Inventory (MBI).
To see whether a one-hour weekly group at work enhances amount of meditation practice. | 8 weeks
  Outcome measured by self-reported average amount of weekly meditation practice.
To see whether a one-hour weekly group at work improves mindfulness. | 8 week
  Outcome measured using Mindful Attention Awareness Scale (MASS) questionnaire.
To see whether a one-hour weekly group at work reduces stress. | 8 weeks
  Outcome measured using the Perceived Stress Scale (PSS10) questionnaire.
To see whether a one-hour weekly group at work decreases burnout. | 8 weeks
  Outcome measured using Maslach Burnout Inventory (MBI) questionnaire.
To see whether a one-hour weekly group at work enhances engagement. | 8 weeks
  Engagement assessed by measuring number of weeks participants actively accessed the intervention website.

SECONDARY OUTCOMES:
Assess if the program is effective at increasing emotional well-being. | 8 weeks, 16 weeks, and 1 year
  Outcome measured using emotional well-being subscale of the RAND Corporation's Medical Outcomes Study Short Form-36 (SF36).
Assess whether the program leads to an increase in work productivity. | 8 weeks, 16 weeks, and 1 year
  Productivity assessed using the call center composite measure of productivity computed monthly for each call service associate.
Assess if the program is effective at increasing vitality. | 8 weeks, 16 weeks, 1 year
  Outcome measured using vitality subscale of the RAND Corporation's Medical Outcomes Study Short Form-36 (SF36).
Assess if the program is effective at increasing emotional role functioning. | 8 weeks, 16 weeks, 1 year
  Outcome measured using emotional role functioning subscale of the RAND Corporation's Medical Outcomes Study Short Form-36 (SF36).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bernstein, MD, Principal Investigator — The Cleveland Clinic; Didier Allexandre, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- See also: Stress Free Now (web-based stress management program) — http://www.clevelandclinicwellness.com/relax